CLINICAL TRIAL: NCT02479841
Title: Health-promoting Competence, Coping and Quality of Life in Patients With COPD
Acronym: REKV-13/1741
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Fonna (Other)
Collaborators: Helse Vest (Other); University of Stavanger (Other)
Responsible Party: Principal Investigator, Heidi B Bringsvor, PhD-candidate, Helse Fonna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HV911836
Record Dates: First submitted 2014-01-22; First posted 2015-06-24 (Estimated); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: COPD; Coping; Quality of Life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Self-Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- self management program (Experimental): Participation in an 11 week self-management program
  Interventions: Other: Self management program
- Control group (No Intervention)

INTERVENTIONS:
Other: Self management program
  Arms: self management program

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a major cause of mortality and disability, and by 2020, it is expected to be the third leading cause of mortality worldwide. COPD is a major public health concern and has considerable impact on health and quality of life.

For this study an evidence based self-management program is developed, the purpose of the study is to see if this self-management program, in collaboration between specialized health services and municipality health services, improves patients with COPD health-promoting competence, coping and quality of life, and reduces health service costs.The study has a RCT design.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD, GOLD 2-4
* Speak and understand norwegian
* Adult

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2015-02; Primary Completion 2017-10 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Change in Health promoting competence, HeiQ | Before, after, and 3,6 and 12 months after comlepting the intervention (self-management program)

CONTACTS AND LOCATIONS:
Overall Officials: Signe B Bentsen, PhDProfessor, Study Director — University of Stavanger, Norway
Locations (1):
- Helse Fonna, Haugesund, Norway